CLINICAL TRIAL: NCT00770458
Title: Non-Invasive Screening for Fetal Aneuploidy: A New Maternal Plasma Marker
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Elizabeth Dragon / Sr. VP Research & Development, Sequenom, Inc.
Other Study IDs: SQNM-Trisomy21-0100
Record Dates: First submitted 2008-10-08; First posted 2008-10-10 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Down Syndrome (Trisomy 21); Edwards Syndrome (Trisomy 18); Patau Syndrome (Trisomy 13); Turner Syndrome
Keywords: Down Syndrome
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women that will undergo standard of care procedures to evaluate fetus for Down Syndrome

SUMMARY:
Validate that circulating cell free fetal nucleic acid can be used to identify a direct marker for fetal aneuploidy, particularly fetal Down Syndrome (DS), that is better than surrogate markers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female
* Subject is pregnant
* Subject is high risk aneuploid patient undergoing genetic counseling, unltrasound screening, amniocentesis and/or CVS procedure
* Subject is willing to provide blood specimen

Exclusion Criteria:

* Subject is not pregnant
* Subject is not willing to provide blood specimen
* Subject is not haveing aneuploid screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fetal care and genetic counseling patients.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Compare investigational assay results for Down Syndrome to standard of care results. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Bombard, MD, Study Director — Sequenom, Inc.
Locations (7):
- United States (7):
  - UCSD Fetal Care & Genetics Center, La Jolla, California
  - San Diego Perinatal Center, San Diego, California
  - Obstetrix Medical Group of San Jose, San Jose, California
  - Obstetrix Medical Group of Colorado, Denver, Colorado
  - Women & Infants, Providence, Rhode Island
  - A.R.U.P., Salt Lake City, Utah
  - Obstetrix Medical Group of Washington, Seattle, Washington